CLINICAL TRIAL: NCT02435056
Title: Continuous Monitoring of Medication Overuse Headache in Europe and Latin America: Development and STAndardization of an Alert and Decision Support System
Brief Title: Medication Overuse Headache (MOH) and an Innovative Approach
Acronym: COMOESTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 215366
Record Dates: First submitted 2015-04-30; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Medication Overuse Headache
Keywords: medication overuse headache; health care system
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classic Approach (No Intervention): Patient fills in a paper diary in order to quantify parameters of MOH (days with headache, acute drugs consumed, etc.)
- IEPR Approach (Experimental): Patient has to use the electronic diary to record days with headache, acute drugs consumed, etc.
  Interventions: Other: IEPR Approach

INTERVENTIONS:
Other: IEPR Approach — Adoption of Interactive Electronic Patient Record (IEPR) that consists of the following clinically-relevant main components:
  * Minimum Data Set for supporting the diagnosis
  * Electronic Diary with associated alerting system for monitoring the patient during the follow-up period
  * Second opinion system for improving the management
  Arms: IEPR Approach

SUMMARY:
Appropriate delivery of quality healthcare requires constant monitoring of the patient during follow up, particularly in the presence of chronic diseases. This approach can be further improved if leading edge tools supporting diagnosis, as well as prediction, identification and monitoring of adverse events are available. COMOESTAS aims to develop an innovative Information Communications Technology (ICT) system that allows patients with a chronic condition to receive continuous and personalized treatment. The whole system is based on an advanced, "all in one" Alerting and Decision Support System that follows patients from the diagnosis and supports the physician in managing the therapy, controlling relevant events impacting on patient safety and activating specific procedures if selected thresholds are exceeded. In the frame of chronic neurological disorders, Medication Overuse Headache (MOH) is a common condition and a major cause of disability. MOH is curable, but its outcome is hampered by a high risk of relapse. It is, therefore, a perfect example of a disorder that can benefit from an ICT-assisted approach developing innovative systems and services for monitoring chronic conditions. COMOESTAS goals will be achieved by improving and integrating the traditional paper headache diaries and calendars into an innovative ICT tool taking into account the complex issues that accompany this peculiar form of headache, which will make the patient a key node in the entire process.

DETAILED DESCRIPTION:
It will be a multicentre parallel group study. The two arms of the clinical protocol will be 1) classic approach to MOH and 2) Interactive Electronic Patient Record (IEPR)-based approach to MOH.

Each arm will last 12 months.

MOH will be diagnosed according to the 2006 MOH-R criteria of the International Headache Society as reported below:

A. Headache present on > 15 days/month.

B. Regular overuse for > 3 months of one or more acute symptomatic drugs:

1. Ergotamine, triptans, opioids or combination analgesic medications on > 10 days/month on a regular basis for > 3 months.
2. Simple analgesics or any combination of ergotamine, triptans, analgesics or opioids on > 15 days/month on a regular basis for >3 months without overuse (> 10 days) of any single class alone.

C. Headache has developed or markedly worsened during medication overuse.

The IEPR approach will be preliminarily tested and validated in small groups of patients during months 6-12 (pilot validation).

Each patient will be evaluated over a period of 7 months.

Classic approach Visit 0: patient is examined and, if suspected to suffer from MOH, is asked to fill in a diary for a month in order to quantify parameters of MOH (days with headache, acute drugs consumed, etc.). Patient has to report that MOH-R criteria were fulfilled for the previous 2 months.

Visit 1: Patient returns to the Centre, diary data are analyzed and recorded, and, if criteria for MOH-R diagnosis are fulfilled and exclusion criteria are ruled out , patient is enrolled in COMOESTAS protocol.

Detoxification: following visit 1, patient undergoes detoxification according to the protocol in Appendix 1. In the subsequent 2 months the patient is instructed to record headache characteristics and consumption of symptomatic drugs on a paper diary.

Visit 2 (2 months after detoxification): patient is visited again; diary is checked; if therapy is successful (patient no longer overuses acute medications for headache) the patient is scheduled for a follow-up visit after 4 months. The patient is asked to keep up recording headache characteristics and consumption of symptomatic drugs on a paper diary for the next 4 months and informed about a telephone contact after 2 months.

Visit 3 (6 months after detoxification): patient is visited again, diary data are collected. Study ends.

IEPR approach Visit 0: patient is examined and, if the minimum data set of the IEPR for MOH is satisfied, the patients is asked to record the headache characteristics as well as acute drugs consumption on a paper diary for a month in order to assess baseline parameters of MOH (days with headache, acute drugs consumed, etc.).

Patient has to report that MOH-R criteria were fulfilled for the previous 2 months.

Visit 1: Patient returns to the Centre, diary data are analyzed and recorded, and, if criteria for MOH diagnosis are confirmed and criteria of exclusion are ruled out, patient is enrolled in COMOESTAS protocol .

Detoxification: following Visit 1, patient undergoes detoxification according to the same protocol adopted for the classic approach. During the detoxification phase, the patient is instructed to use the electronic diary and is then asked to fill the electronic diary on a regular basis (preferably daily or at least weekly) for the next 6 months.

Visit 2 (2 months after detoxification): patient is visited again; if therapy is successful (patient no longer overuses acute medications for headache), MOH diagnosis the patient is scheduled for a follow-up visit after 4 months and informed about a telephone contact after 2 months. The patient is asked to keep up filling the electronic diary for the next 4 months.

Visit 3: the patient is visited again. Study ends.

ELIGIBILITY:
Inclusion Criteria:

Patients with MOH

Exclusion Criteria:

1. a current diagnosis of co-existent, significant and complicating medical or psychiatric illnesses
2. significant overuse of "pure" opioids (patients overusing combination drugs containing opioids are allowed), benzodiazepines, and barbiturates,
3. overuse of alcohol and other drugs of addiction,
4. current treatment with migraine prophylactic drugs
5. inefficacy of previous adequate detoxification programmes
6. inability to provide reliable information about medical history
7. pregnancy or breast feeding
8. inability to learn how to use paper or electronic diaries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Relapse Rate Follow up | 6 month
  Relapse Rate 6 months after withdrawal of patients with medication overuse. Relapse will be defined as use of ergotamine, triptans, opioids or combination analgesic medications on > 10 days/month or use of simple analgesics or any combination of ergotamine, triptans, analgesics or opioids on > 15 days/month during the previous month, with the exclusion of month +1.

SECONDARY OUTCOMES:
Days with headache | 6 month
  Number of days with headache before and after detoxification in the two arms (month -1 vs. month +6)
Days per month with migraine | 6 month
  Number of days per month with migraine before and after detoxification in the two arms (month -1 vs. month +6)
MOH patients/total number of headache | 12 month
  Number of MOH patients/total number of headache patients during the recruitment period (6-12 months ) of the two arms
MOH patients/total number of headache | 24 month
  Number of MOH patients/total number of headache patients during the recruitment period (18-24 months ) of the two arms
Drop-outs | 24 month
  Number of drop-outs in the two arms
Midas scores | 24 month
  Changes in Midas scores in the two arms
HURT scores | 24 month
  Changes in HURT scores in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Nappi, MD, Study Director — IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia, ITALY; Rigmor Jensen, MD, PhD, Principal Investigator — Glostrup Hospital, Copenaghen, Denmark; Zaza Katsarava, MD, PHD, MSc, Principal Investigator — Universitaetsklinikum, Essen, Germany; Jorge Leston, MD, Principal Investigator — Fundacion para la Lucha contra las Enfermedades Neurologicas de la Infancia, Argentina; Ricardo Fadic, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Miguel JA Lainez, MD, PhD, Principal Investigator — Fundacion de la Comunidad Valenciana para la Investigacion Biomedica, la Docencia Y la Cooperacion Internacional y para el Desarrollo del Hospital Clinico Universitario De Valencia, Spain; Marco Pagani, Manager, Principal Investigator — Consorzio di Bioingegneria Medica, Pavia, Italy; Nestor Gorini, Principal Investigator — Ministerio de la Salud de la Provincia de Buenos Aires, Argentina; Santiago Spadafora, Principal Investigator — Fundacion Isalud, Buenos Aires, Argentina

REFERENCES:
- [Background] Rossi P, Di Lorenzo C, Faroni J, Cesarino F, Nappi G. Advice alone vs. structured detoxification programmes for medication overuse headache: a prospective, randomized, open-label trial in transformed migraine patients with low medical needs. Cephalalgia. 2006 Sep;26(9):1097-105. doi: 10.1111/j.1468-2982.2006.01175.x. PMID 16919060
- [Background] Diener HC, Limmroth V. Medication-overuse headache: a worldwide problem. Lancet Neurol. 2004 Aug;3(8):475-83. doi: 10.1016/S1474-4422(04)00824-5. PMID 15261608
- [Background] Zeeberg P, Olesen J, Jensen R. Discontinuation of medication overuse in headache patients: recovery of therapeutic responsiveness. Cephalalgia. 2006 Oct;26(10):1192-8. doi: 10.1111/j.1468-2982.2006.01190.x. PMID 16961785
- [Background] Zeeberg P, Olesen J, Jensen R. Probable medication-overuse headache: the effect of a 2-month drug-free period. Neurology. 2006 Jun 27;66(12):1894-8. doi: 10.1212/01.wnl.0000217914.30994.bd. Epub 2006 May 17. PMID 16707727
- [Background] Haag G, Baar H, Grotemeyer KH, Pfaffenrath V, Ribbat MJ, Diener HC. [Prophylaxis and treatment of drug-induced persistent headache. Therapy recommendation of the German Society for Migraine and Headache]. Schmerz. 1999 Feb 18;13(1):52-7. doi: 10.1007/s004829900016. No abstract available. German. PMID 12799950
- [Background] Headache Classification Committee; Olesen J, Bousser MG, Diener HC, Dodick D, First M, Goadsby PJ, Gobel H, Lainez MJ, Lance JW, Lipton RB, Nappi G, Sakai F, Schoenen J, Silberstein SD, Steiner TJ. New appendix criteria open for a broader concept of chronic migraine. Cephalalgia. 2006 Jun;26(6):742-6. doi: 10.1111/j.1468-2982.2006.01172.x. PMID 16686915
- [Derived] Jellestad PL, Carlsen LN, Westergaard ML, Munksgaard SB, Bendtsen L, Lainez M, Fadic R, Katsarava Z, Goicochea MT, Spadafora S, Jensen RH, Nappi G, Tassorelli C; COMOESTAS Consortium. Economic benefits of treating medication-overuse headache - results from the multicenter COMOESTAS project. Cephalalgia. 2019 Feb;39(2):274-285. doi: 10.1177/0333102418786265. Epub 2018 Jul 8. PMID 29984608
- [Derived] Tassorelli C, Jensen R, Allena M, De Icco R, Katsarava Z, Miguel Lainez J, Leston JA, Fadic R, Spadafora S, Pagani M, Nappi G; COMOESTAS Consortium. The added value of an electronic monitoring and alerting system in the management of medication-overuse headache: A controlled multicentre study. Cephalalgia. 2017 Oct;37(12):1115-1125. doi: 10.1177/0333102416660549. Epub 2016 Jul 20. PMID 27440251